CLINICAL TRIAL: NCT03159689
Title: Mixed Nuts as Healthy Snack: Effect on Body Weight and Composition
Brief Title: The Effect of a Healthy Snack on Body Weight and Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-000361
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed Tree Nuts (Experimental): a hypo caloric weight loss dietary plan with mixed tree nuts
  Interventions: Other: Mixed Tree Nuts
- Pretzels (Active Comparator): a hypo caloric weight loss dietary plan with pretzels
  Interventions: Other: Pretzels

INTERVENTIONS:
Other: Mixed Tree Nuts — Individuals on a hypo caloric weight loss dietary plan supplemented with 1.5oz mixed tree nuts
  Arms: Mixed Tree Nuts
Other: Pretzels — Individuals on a hypo caloric weight loss dietary plan supplemented with 1.5oz pretzels
  Arms: Pretzels

SUMMARY:
The results from this study may help to explain if incorporating mixed nuts in a reduced calorie diet will lead to weight loss.

DETAILED DESCRIPTION:
This study will compare two energy reduced diets; one diet will include one serving of mixed nuts (1.5oz) per day, while the other diet will include an equal amount of calories from a carbohydrate source, such as a pretzel snack. All subjects will receive a dietary plan that reduces their usual intake by 500kcal/day with the same percentage of fat, protein and carbohydrates for the first 12 weeks followed a diet with their usual intake for 12 weeks without nuts or pretzels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 40-60 years of age (female premenopausal).
* Body Mass Index (BMI) 27.0-35.0 kg/m2.
* Not currently taking a prescription or over the counter medication for weight loss.
* Not currently enrolled in any commercial weight loss program (e.g. Jenny Craig, Weight Watchers), internet based weight-management program, self-help group (e.g. Overeaters Anonymous) or participating in any food preparation/delivery program. If subject is willing to discontinue program immediately and willing to refrain from program for duration of study, he/she may be included after a two-week washout period.
* Willing to keep and turn in a daily log/compliance book as required by study protocol.
* Willingness and ability to make all scheduled appointments.
* Willing to follow dietary recommendations required by study protocol.
* Willingness to periodically have small blood samples drawn as indicated in the protocol.

Exclusion Criteria:

* More than a 5-pound weight gain or weight loss within the 3 months prior to enrollment in the study.
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* History of Type I or Type II diabetes, major surgery, heart problems (e.g. angina, bypass surgery, MI, etc.), presence of implanted cardiac defibrillator or pacemaker, uncontrolled hypertension/high blood pressure, gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease, inflammatory bowel disease, fatty liver or cancer within three months of enrollment
* History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy).
* Following a diet that requires the elimination of FODMAPS (Fermentable Oligosaccharides, Disaccharides, Monosaccharides And Polyols)
* Following a specific diet that restricts specific food groups (eg. Paleo) or with extreme macronutrient ratios (carbohydrates, fats and proteins).
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia nervosa or binge eating disorder.
* Women who are pregnant, lactating or trying to become pregnant.
* Currently taking any prescription medication for less than 3 months.
* Currently taking any prescriptions drugs or supplements that may impact weight regulation
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and/or unwilling to limit intake to less than 3 drinks per week during study participation or history of alcohol dependency.
* Known allergy to almond, pistachio, walnut, macadamia, cashews, hazelnuts, or pecan nuts.
* Participation in another clinical trial within 30 days prior to enrollment.
* Currently smoking cigarettes.
* Any known clinically significant food allergy or intolerance.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | baseline to Week 24
  Weight loss as determined by body composition and body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, 900 Veteran Avenue, WH 14-187, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD